CLINICAL TRIAL: NCT01887717
Title: A Prospective Randomized Clinical Trial on 90Yttrium Trans-arterial Radio-Embolization (TheraSphere®) vs. Standard of Care (Sorafenib) for the Treatment of Advanced Hepatocellular Carcinoma (HCC) With Portal Vein Thrombosis (PVT)
Brief Title: Efficacy Evaluation of TheraSphere to Treat Inoperable Liver Cancer With Blockage of the Portal Vein
Acronym: YES-P
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor Accrual.
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS-104; 2012-005375-14 (EudraCT Number)
Record Dates: First submitted 2013-06-03; First posted 2013-06-27 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; portal vein thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TheraSphere (Experimental): Participants will receive TheraSphere at a dose consistent with the approved product label to the treated lobe of the liver. TheraSphere will be administered through the hepatic artery. The target dose will be 120 Gy + 10%. Dose reduction to a minimum dose of 80 Gy + 10% will be permitted to manage radiation exposure to the lungs. Re-treatment of the same participant/lobe with further cycles of TheraSphere will be permitted if a treatable progression is detected during follow-up evaluations. Any re-treatment will take place at least 28 days after the previous TheraSphere treatment administered to that lobe. Participants can receive a subsequent TheraSphere administration in the absence of radiological progression criteria at the Investigator's discretion. A maximum of 3 TheraSphere administrations will be permitted.
  Interventions: Device: TheraSphere®
- Sorafenib (Active Comparator): Participants will receive sorafenib, oral tablets, 400 milligrams (mg) twice daily in accordance with the package insert. Treatment is to continue until the participant is no longer clinically benefiting from therapy or until unacceptable toxicity occurs. Medically appropriate dose adjustments and drug holidays due to adverse events (AEs) and toxicity will be allowed.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Device: TheraSphere® — Intrahepatic treatment of advanced hepatocellular carcinoma
  Other Names: yttrium-90 microspheres
  Arms: TheraSphere
Drug: Sorafenib — Standard of care therapy for treatment of advanced hepatocellular carcinoma
  Other Names: Nexavar®
  Arms: Sorafenib

SUMMARY:
This is a two-arm, open-label, prospective, multi-center, randomized, active-controlled clinical trial to assess efficacy and safety of TheraSphere in comparison to standard of care therapy (sorafenib) in the treatment of participants with inoperable liver cancer and blockage of the portal vein.

DETAILED DESCRIPTION:
The objective of this Phase III, prospective randomized trial is to determine whether TheraSphere provides a meaningful benefit in survival in comparison with the standard of care (sorafenib) in participants with good hepatic function and advanced hepatocellular carcinoma (HCC) associated with portal vein thrombosis (PVT).

This is an open-label prospective, multi-center, randomized, controlled clinical trial that will evaluate the use of TheraSphere compared to standard-of-care sorafenib alone.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 years of age, regardless of race or gender
* Advanced unresectable hepatocellular carcinoma with branch portal vein thrombosis (confirmed by non-invasive criteria European Association for the Study of the Liver [EASL]/American Association for the Study of Liver Diseases [AASLD], mandatory by histology in non-cirrhotic participants); can be naive or recurrent HCC after curative treatment ( >6 months before randomization)
* Unilobar disease
* Child Pugh A
* Tumor volume ≤70% of liver volume (determined by visual estimation)
* At least one uni-dimensional HCC target lesion assessable by computed tomography (CT) or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Platelets ≥ 50*10^3/microliter (µL)
* White blood cell (WBC) ≥1.5*10^3/microliter (µL)
* Aspartate transaminase (AST)/ alanine aminotransferase (ALT) ≤5 times upper limit of normal
* Creatinine ≤2.0 mg/deciliter (dL)
* Life expectancy >3 months
* Signed informed consent

Exclusion Criteria:

* Confirmed extra hepatic metastases. Participants with indeterminate hepatic hilar lymph nodes up to 2.5 centimeters (cm) in greatest dimension, or with indeterminate lung nodules (single lesion between 1-1.5 cm, or multiple smaller lesions with a total diameter of ≤2 cm) may be included if metastatic disease is deemed unlikely
* Known contraindication to standard-of-care sorafenib including allergic reaction, pill swallowing difficulty, uncontrolled hypertension or history of cardiac disease, significant GI bleed within 30 days, and renal failure including dialysis
* Evidence of hepatic vein invasion or caval thrombosis
* Evidence of chronic obstructive pulmonary disease
* Indication for any possible curative treatment after multidisciplinary assessment (surgery, ablation, transplantation)
* Previous treatment with sorafenib for more than 4 weeks during the previous 2 months; prior sorafenib-related toxicity
* Initiation of anti-tumor therapy including chemotherapy or investigational drug treatment within 30 days before beginning study
* Prior transarterial chemoembolization (TACE) <6 months prior to screening phase in case of participants progressing from an intermediate to an advanced stage due to occurrence of PVT
* On a transplant list
* History of organ allograft
* Contraindications to angiography or selective visceral catheterization
* History of severe allergy or intolerance to contrast agents, narcotics, sedatives, or atropine that cannot be managed medically
* Prior external beam radiation therapy to the liver
* Evidence of continuing adverse effect of prior therapy
* Active gastrointestinal (GI) bleeding and any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents
* Evidence of any disease or condition that would place the participant at undue risk and preclude safe use of TheraSphere treatment
* Females of child-bearing potential must have a negative serum test
* No participation in concurrent clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02-27 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, Principal Investigator — Istituto Tumori Nazionale, Milan, Italy; Riad Salem, MD, Principal Investigator — Northwestern University Chicago Illinois
Locations (19):
- United States (2):
  - Northwestern Medical Faculty Foundation, Div of Hematology/Oncology, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Paoli-Calmettes Institute, Marseille, France
- Italy (9):
  - UO Radiologia, Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ASO-Santa Croce e Carle di Cuneo, Cuneo
  - Fondazione IRCCS Ca Grande, Milan
  - S.C Radiologia Interventistica, A.O.Ospedale Niguarda Ca Granda, Milan
  - Fondazione Istituto Nazionale Tumori di Milano, Milan
  - Azienda Ospedaliera Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - University of Pisa, Pisa
  - Policlinico A. Gemelli, Rome
- Spain (4):
  - Hospital Clínic Barcelona. IDIBAPS. CIBEREHD. Liver Unit, Barcelona
  - Bulevar Sur s/n, Madrid
  - Hospital Universitario Puerta de Hierro, Gastroenterology & Hepatology Dept, Madrid
  - Hospital Universitari i Politecnic la Fe, Valencia
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Free London NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment started on February 27, 2014 and was terminated prematurely on March 31, 2016 due to slow recruitment, after randomization of 36 participants. Participants were enrolled at 13 centers in 6 countries (United States, Belgium, Spain, France, England, and Italy).
Pre-assignment Details: Participants were randomized 1:1 to the TheraSphere group or control group. To balance the treatment groups, participants were stratified at randomization on the basis of serum level of alpha-fetoprotein (AFP) (<400 nanograms/milliliter [ng/mL] versus >400 ng/mL) and study center.
Groups:
- TheraSphere: Participants received TheraSphere at a dose consistent with the approved package insert to the treated lobe of the liver. TheraSphere was administered through the hepatic artery. The targeted dose was 120 Gy + 10%. Dose reduction to a minimum dose of 80 Gy + 10% was permitted to manage radiation exposure to the lungs. Re-treatment of the same participant/lobe with further cycles of TheraSphere was permitted if a treatable progression was detected during follow-up evaluations. Any re-treatment took place at least 28 days after the previous TheraSphere treatment administered to that lobe. Participants could receive a subsequent TheraSphere administration in the absence of radiological progression criteria at the Investigator's discretion. A maximum of 3 TheraSphere administrations was permitted.
- Sorafenib: Participants received sorafenib, oral tablets, 400 milligrams (mg) twice daily in accordance with the package insert. Treatment was to continue until the participant was no longer clinically benefiting from therapy or until unacceptable toxicity occurred. Medically appropriate dose adjustments and drug holidays due to adverse events (AEs) and toxicity were allowed.
Period: Overall Study
Arm/Group | TheraSphere | Sorafenib
Started | 17 | 19
Received at Least 1 Dose of Study Drug | 15 | 16
Completed | 11 | 8
Not Completed | 6 | 11
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Physician Decision | 0 | 2
Not completed — Administrative reasons | 5 | 2

BASELINE CHARACTERISTICS:
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Groups:
- Total: Total of all reporting groups
Arm/Group | TheraSphere | Sorafenib | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (8.39) | 64.4 (8.73) | 65.8 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
AFP [Mean (Standard Deviation); unit: ng/mL] | 3260.6 (10846.39) | 5365.6 (15538.93) | 4347.1 (13295.61)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) From Time of Randomization
Description: OS was calculated as the interval between the randomization date and the date of death for any cause, with censoring at the date of last contact for participants alive.
Time Frame: Randomization up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Median (Full Range); unit: months
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
months | 14.5 [2.3 to 22.0] | 18.2 [2.9 to 18.2]

2. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from randomization until date of first radiological progression (including new liver lesions and extra-hepatic lesions) separately according to Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1 criteria, modified RECIST (mRECIST) criteria, and European Association for the Study of the Liver (EASL) criteria (assessed bi-dimensionally on enhancing tissue) as assessed by Investigator determination. Progression was defined as an increase >25% in the size of ≥1 measurable lesions (EASL) and ≥20% increase in the sum of the diameter of viable of target lesion (mRECIST). RECIST v1.1 categorized new lesions as Progressive Disease. TTP (Months)=(Date of event/censor - Date of Randomization + 1)/ 30.4375.
Time Frame: Randomization up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Median (Full Range); unit: months
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
months
  RECIST 1.1 Criteria | 6.2 [1.6 to 18.7] | 3.7 [1.6 to 29.2]
  mRECIST Criteria | 17.0 [1.6 to 18.7] | 4.1 [1.6 to 29.2]
  EASL Criteria | 8.1 [1.6 to 18.7] | 3.5 [1.6 to 5.5]

3. Secondary Outcome: Time to Worsening Portal Vein Thrombosis (PVT)
Description: Time of randomization to time of any change in classification of PVT type by ≥1 sub-type based on Investigator assessment. At screening and every 8 weeks after, PVT categorized based on dynamic imaging studies as: Type I: segmental, in ≥1 of 8 branches of the portal vein; Type II: branched, left or right branches of the portal vein; Type III: modified on the basis of extension of the tumor thrombus; Type IIIa: eligible for study, thrombus involving the main trunk, allowing blood flow to contralateral lobe (no thrombosis); Type IIIb: NOT eligible for study, thrombus in the main portal trunk occluding blood flow to contralateral lobe; and Type IV: main PVT, NOT eligible for study, extended (mesenteric or splenic veins and/or sovra-hepatic veins). Time to Worsening of PVT (Months)=(Date of event/censor-Date of Randomization+1)/30.4375. Median time to event defined as time it is expected for half of the participants to experience the event. Data analyzed using the Kaplan-Meier method.
Time Frame: Baseline (Randomization) up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
months | 8.2 [5.7 to NA] — NA=Not available. Too few participants experienced the event to estimate the upper limit using the Kaplan-Meier method. | NA [1.9 to NA] — Too few participants experienced the event to estimate the median and upper limit using the Kaplan-Meier method.

4. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Description: TTSP calculated as interval between randomization and symptomatic progression. Symptomatic progression defined as clinical progress to Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≥2 with or without tumor progression on imaging. Deterioration in PS was confirmed at the evaluation 8 weeks later. First date at which ECOG performance status was ≥2 was used as end date in TTSP analysis (assuming next subsequent visit confirmed deterioration). TTSP (Months)=(Date of ECOG >2-Date of Randomization+1)/30.4375. ECOG PS Scale: 0=Asymptomatic and fully active; 1=Symptomatic, fully ambulatory, restricted in physically strenuous activity; 2=Symptomatic, ambulatory, capable of self-care, more than 50% of waking hours are spent out of bed; 4=Completely disabled, no self-care, bedridden. Median time to event defined as time it is expected for half of the participants to experience the event. Data analyzed using the Kaplan-Meier method.
Time Frame: Randomization up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Median (Full Range); unit: months
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
months | NA [20.3 to NA] — Too few participants experienced the event to estimate the median and upper limit using the Kaplan-Meier method. | NA [NA to NA] — Too few participants experienced the event to estimate the median, lower limit, and upper limit using the Kaplan-Meier method.

5. Secondary Outcome: Number of Participants With Tumor Response
Description: Tumor Response was based on the radiological tumor assessment and was categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Tumor response was assessed using RECIST version (v) 1.1, mRECIST, and EASL criteria. Criteria included: CR=disappearance of all enhanced tumor areas (EASL) and disappearance of any intratumoral arterial enhancement in all target lesions (mRECIST); PR= decrease >50% of enhanced areas (EASL) and ≥30% decrease in the sum of diameters of viable target lesions (mRECIST); SD=neither CR, PR, PD (EASL/mRECIST); PD=an increase >25% in the size of ≥1 measurable lesions (EASL) and ≥20% increase in the sum of the diameter of viable of target lesion (mRECIST). RECIST v 1.1 categorized new lesions as Progressive Disease only and the non-target lesions needed to have no progressive disease to be categorized as CR or PR. One month=30.4375 days.
Time Frame: Baseline up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib and with available Tumor Response data.
Measure: Count of Participants; unit: Participants
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
Participants
  RECIST CR | 0 | 0
  RECIST PR | 1 | 0
  mRECIST CR | 0 | 0
  mRECIST PR | 1 | 0
  EASL CR | 0 | 0
  EASL PR | 0 | 0

6. Secondary Outcome: Change From Baseline in Quality of Life (QoL) as Assessed by the FACT-Hep Questionnaire
Description: The Functional Assessment Cancer of Therapy-Hepatobiliary (FACT-Hep) Questionnaire uses participant reported outcome (PRO) scores. The FACT-Hep Trial Outcome Index (TOI) is the sum of the subscales scores in Personal Well-Being (PWB), Functional Well-Being (FWB), and Hepatobiliary Cancer Subscale (HCS). The higher the score, the better the QoL, with a range 0-128. Baseline data and change from Baseline data is presented.
Time Frame: Baseline (Randomization), participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib and with evaluable TOI data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 13 | 14
score on a scale
  Baseline TOI | 94.63 (16.692) | 103.54 (14.934)
  Month 30 TOI: number analyzed (Participants) | 1 | 0
  Month 30 TOI | -5.20 (NA) — Standard deviation cannot be calculated with an N of 1. |

7. Secondary Outcome: Time to Deterioration QoL (TTDQoL)
Description: TTDQoL was calculated as the interval between the randomization date and deterioration in QoL. The FACT-Hep Questionnaire uses PRO scores. A deterioration in QoL is defined as a >7-point decline in the total score or death, whichever occurred first. The FACT-Hep Total Score is the sum of the subscales scores in PWB, Social/Family Well-Being (SWB), Emotional Well-Being (EWB), FWB, and HCS. The higher the score, the better the QoL, with a range 0-180. TTDQoL (Months)=(Date of change from baseline in FACT-Hep ≥7 or death) - Date of Randomization + 1.
Time Frame: Baseline (Randomization) up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Mean (Full Range); unit: months
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
months | 2.5 [0.6 to 24.0] | 1.6 [0.9 to 9.0]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An TEAE is any untoward medical occurrence or undesirable event(s) experienced in a participant that begins or worsens following administration of the study drug or study treatment, whether or not considered related to the treatment by the Investigator. A serious adverse event (SAE) was an adverse event (AE) resulting in any of the following outcomes or deemed significant for any other reason, death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, or congenital anomaly. AEs included both SAEs and non-serious AEs. AEs were classified according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 (CTCAE) and coded using the Medical Dictionary for Regulatory Activities (MedDRA). A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Randomization up to participant's death (maximum time = up to Month 30)
Population: Participants who received at least 1 dose of TheraSphere or Sorafenib.
Measure: Count of Participants; unit: Participants
Arm/Group | TheraSphere | Sorafenib
Number analyzed (Participants) | 15 | 16
Participants
  TEAE | 6 | 16
  Adverse Device Event (ADE) | 3 | 0
  Angiographic Related TEAE | 3 | 0
  TEAE CTCAE ≥ Grade 3 | 1 | 9
  Treatment Emergent SAE | 0 | 7
  Related Serious Adverse Device Effect (SADE) | 0 | 0
  TEAE with an Outcome of Death | 0 | 4
  TEAE with Action Taken of Sorafenib Discontinued | 0 | 2

ADVERSE EVENTS:
Time Frame: Randomization up to participant's death (maximum time = up to Month 30)
Arm/Group | TheraSphere | Sorafenib
All-Cause Mortality (participants affected / at risk) | 15/15 | 16/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 12/16
Other Adverse Events (participants affected / at risk) | 6/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TheraSphere (N=15) | Sorafenib (N=16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
General Physical Health Deterioration (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | TheraSphere (N=15) | Sorafenib (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 7
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Steatorrhoea (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 2 | 5
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
General physical health deterioration (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 4
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 2
Eosinophil count decreased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 3
Memory impairment (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0/12 | 1/13 — This is a sex-specific adverse event that only affects male participants.
Scrotal erythema (Reproductive system and breast disorders) | 0/12 | 1/13 — This is a sex-specific adverse event that only affects male participants.
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Hyperaemia (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 3
Peripheral coldness (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
On 23 May 2017, the Sponsor announced early termination of the study because fewer than half of the participants remained in follow-up resulting in to few participants for the study to be continued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BTG can require Investigator to postpone publications/presentations for up to 12 months so data from all sites can be published. BTG will limit review of Investigator's draft to confirm Confidential Information is not being disclosed. If BTG notes publishing Study results may affect obtaining a patent, Investigator will not publish for up to 60 days until patent application is filed. Investigator will acknowledge BTG in any publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2014-08-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT01887717/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT01887717/SAP_001.pdf